CLINICAL TRIAL: NCT01577667
Title: Comparative Monocenter RCT Comparing Safety and Efficacy of an Automated Closed-loop Oxygenation and Ventilation(IntelliVent® System - HAMILTON MEDICAL AG) With Non-automated Conventional Ventilation and Oxygenation
Brief Title: Intellivent Versus Conventional Ventilation
Acronym: Intellivent
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Medical AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Intellivent RCT1
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Respiratory Failure; Self Efficacy
Keywords: automation; closed loop; oxygenation; ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional ventilation (No Intervention): Usual ventilation is administered according to the protocols implemented in the unit
- Intellivent (Experimental): Intellivent is a ventilatory mode included in ventilator S1, Hamilton Medical. Intervention: the patient is ventilated with the same ventilator than in the conventionnal group; but the "ASV-Intellivent" ventilation has to be activated via a dedicated key on the ventilator screen.
  IntelliVent® activation requires selecting the kind of patient: ARDS, COPD and whether hemodynamic instability exists.
  The initial settings are IntelliVent® by default settings (% MV: 110%, PEEP: 5 cm H2O, FiO2: 60% - 100% in case of ARDS).
  Therefore modification of these various parameters is automatic. FiO2 and PEP are modified according to SpO2; %MV according to EtCO2.
  Interventions: Device: Intellivent; automatic mode implemented on a S1 ventilator

INTERVENTIONS:
Device: Intellivent; automatic mode implemented on a S1 ventilator — Intellivent allows an automatic adjustment of the following parameters: FiO2, PEEP and %VM according to adjusted parameters: Size, SpO2 and EtCO2
  Other Names: Closed-loop ventilation
  Arms: Intellivent

SUMMARY:
Partial automation of mechanical ventilation in resuscitation has been available for several years. New modalities are being developed to completely automate ventilation and oxygenation parameters (IntelliVent®.

This pilot study compares over a 48h period the safety and efficacy of IntelliVent®, versus a conventional ventilation modality.

DETAILED DESCRIPTION:
Rational: Partial automation of mechanical ventilation in resuscitation has been available for several years. It can deliver a continuous ventilation adapted in real time to the patient's clinical condition,and decrease care workload and ventilation weaning duration. New modalities are being developed to completely automate ventilation and oxygenation parameters (IntelliVent®) and preliminary studies show that over short periods (2 to 4 h) such a system can ventilate patients more optimally and more safely, with a better ventilation efficiency (comparable effect on gas exchanges for a less "aggressive" ventilation). This pilot study compares over a longer period (48 hours), the safety and efficacy of IntelliVent®, versus a usual ventilation modality.

Type of study: Monocenter, comparative, prospective, randomized, parallel study.

Objective: To assess IntelliVent® safety, efficacy, and care workload.

Assessment criteria:

* Safety is assessed by measuring the number of times it is necessary to manually intervene on the ventilator settings because for one the following parameters: A range SpO2, EtCO2, plateau pressure (Pplat), tidal volume (VT), respiratory rate (RR),values considered as non-optimal, as defined a priori and consensually by a panel of experts.
* Efficacy, in terms of ventilation, is assessed by the time spent within a range EtCO2 and Pplat and VT and RR values considered as optimal, as defined a priori and consensually by a panel of experts.

Efficacy, in terms of oxygenation, is assessed by the time spent within a range SpO2 values considered as optimal, as defined a priori and consensually by a panel of experts.

- Care workload is assessed by the number of ventilator setting adjustments by nursing staff in each group.

Number of subjects: 80 patients receiving invasive mechanical ventilation for acute respiratory failure.

Methods: The selected patients presenting with inclusion criteria are ventilated either with IntelliVent® or with the unit's usual ventilation following a random selection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient under invasive ventilation for more than 6 hours and for a planned duration of at least 48 hours
* Body Mass Index (current weight (kg)/height (m)²) < 40
* Signature of an informed consent by the family

Exclusion Criteria:

* Need for ventricular assistance with intra-aortic balloon counterpulsation.
* Presence of a bronchopleural fistula
* Pregnant women: A pregnancy blood test will be performed in women of reproductive age. The results will be communicated to the patient by a physician of her choice.
* Adults under guardianship
* People deprived of freedom
* Inclusion in another study protocol under consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety | 48 Hours
  Safety is assessed by measuring the number of times it is necessary to manually intervene on the ventilator settings because for one the following parameters: A range SpO2, EtCO2, plateau pressure (Pplat), tidal volume (VT), respiratory rate (RR) values considered as non-optimal, as defined a priori and consensually by a panel of experts.

SECONDARY OUTCOMES:
Efficacy | 48 Hours
  Efficacy, in terms of ventilation, is assessed by the time spent within a range EtCO2 and Pplat-proxi and VT and RR values considered as optimal, as defined a priori and consensually by a panel of experts.
  Efficacy, in terms of oxygenation, is assessed by the time spent within a range SpO2 values considered as optimal, as defined a priori and consensually by a panel of experts.
Care workload | 48H
  Care workload is assessed by the number of ventilator setting adjustments by nursing staff in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François Laterre, Pr, Principal Investigator — Reanimation, Cliniques Universitaires Saint Luc
Locations (1):
- Polyvalent Intensive Care, St Luc Clinics, Brussels, Belgium